CLINICAL TRIAL: NCT04677881
Title: Health Effects and Consumer Aspects of Different Types of Bread
Brief Title: Health Effects of Different Types of Bread
Acronym: HELFAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: University of Oslo (Other); Mesterbakeren (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 96264
Record Dates: First submitted 2020-11-26; First posted 2020-12-21 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2020-10

CONDITIONS: IBS

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wholegrain bread with yeast (Placebo Comparator): The control group will be given min. 5 slices of bread baked with yeast per day.
  Interventions: Other: Intervention group
- Wholegrain bread with sourdough (Experimental): The experimental group will be given min. 5 slices of bread baked with sourdough per day.
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: Intervention group — intervention group: bread with sourdough control group: bread with yeast

SUMMARY:
Dietary fiber is well known to have health promoting effects, including reduced blood glucose and cholesterol levels. Bread is the most important source of dietary fiber in the Norwegian diet. Production of bread has changed from the traditionally use of sourdough, to yeast (Saccharomyces cerevisiae) as the dominating leavening agent in modern industrial production. Sourdough naturally contains bacteria, and through the fermentation process these bacteria release several components that are not found in modern bread using yeast. It has been shown that sourdough may have positive health effects, including on blood glucose regulation. The aim of the project is to investigate if intake of sourdough may give positive health effects compared to beard with yeast.

DETAILED DESCRIPTION:
The investigators aim to include approximately 20 participants in this randomized controlled double-blind cross-over study lasting for 5 weeks.

All participants will be given bread baked with yeast for a 2 weeks run-in period. The participants will then be randomly assigned to either 1 week intervention with bread baked with yeast or sourdough, before a 1 week wash-out period with yeast bread. During the last 1 week intervention period the participants starting with bread baked with yeast will be given sourdough and vice versa.

Questionnaires (GSRS-IBS, BSC, FFQ), blood samples, and feces samples will be collected before and after the intervention periods.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults who restrict their intake of bread due to stomach ache.

Exclusion Criteria:

* Chronic metabolic diseases, such as diabetes type 1 or 2, cardiovascular diseases and cancer last 6 months
* Gut diseases, including Chron's disease, ulcers colitis
* Food allergies or intolerance
* Pregnant and/or lactating
* Smokers
* BMI <18,5 and >27 kg/m2
* Planed weight reduction and/or ± 5% weight change last 3 months
* Blood donor last 2 months and during the study period
* Not willing to quit taking dietary supplements, including probiotics, cod liver oil etc., 4 weeks prior to study start and during the study
* Use of antibiotics <3 months prior to study start and during the study
* Alcohol intake >40 g/day
* Hormone treatment (except contraceptives)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale-irritable bowl syndrome (GSRS-IBS) | 5 weeks
  GSRS-IBS analysis after intervention with bread baked with yeast versus sourdough with the following response scale: 1 (no discomfort at all) to 7 (very severe discomfort)

SECONDARY OUTCOMES:
Bristol stool chart (BSC) | 5 weeks
  BSC analyses after intervention with bread baked with yeast versus sourdough with a scale from 1 (separate hard lumps, like nuts) to 7 (watery, no solid pieces)
Blood C-peptide, total cholesterol, triglycerides, fatty acid profile, and short chain fatty acids | 5 weeks
  Blood analyses of C-peptide, total cholesterol, triglycerides, fatty acid profile, and short chain fatty acids after intervention with bread baked with yeast versus sourdough
Feces microbiota analysis performed with Bio-Me's Precision Microbiome Profiling platform (PMP™) | 5 weeks
  Feces analyses of microbiota after intervention with bread baked with yeast versus sourdough
Iron, selenium and zinc in blood | 5 weeks
  Blood analysis of iron, selenium and zinc after intervention with bread baked with yeast versus sourdough

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Telle-Hansen, PhD, Principal Investigator — Oslo and Akershus University College
Locations (1):
- Vibeke Telle-Hansen, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No